CLINICAL TRIAL: NCT05321459
Title: New Predictive Tool of Awakening in Comatose Patients in the Intensive Care Unit
Brief Title: Predictive Outcome in Comatose Patients
Acronym: PRECOM
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ecole Normale Supérieure de Paris (Unknown)
Responsible Party: Sponsor
Other Study IDs: AOR 20045
Record Dates: First submitted 2022-03-14; First posted 2022-04-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Coma; Heart Arrest; Cardiopulmonary Resuscitation
Keywords: Post cardiac arrest for comatose patients; Electroencephalography; Somatosensory evoked potentials; Auditory evoked potentials; Prognosis; Algorithms; Classification
MeSH Terms: conditions — Coma; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Comatose patients in intensive care unit: Patient admitted in the intensive care unit (ICU) for post cardiac arrest (CA) coma, persistent for at least 3 days after CA.
  Interventions: Other: Neurological prognosis

INTERVENTIONS:
Other: Neurological prognosis — In usual practice, in intensive care unit, evaluating the neurological prognosis of comatose patients after cardiac arrest requires a multimodal approach combining standardized clinical examination, serum biomarkers, imaging and classically electrophysiological examinations (among them auditive evoked potentials or AEP).
  An algorithm (PRECOM tool) which has been previously developed from the signal extracted from AEP allows to visually classify the patients after processing signal by the algorithm in a cluster of points with a high specificity into "good neurological prognosis" and "bad neurological prognosis".
  The AEP signals recorded in the 1st and 2nd week of patient inclusion are to be collected by the neurophysiologist. At the end of the patient's participation in the study, these data will be encrypted, anonymized and transmitted to the mathematician to be processed by the PRECOM tool.

SUMMARY:
Evaluating the prognosis of comatose patients after cardiac arrest (CA) in the intensive care unit (ICU) remains challenging. It requires a multimodal approach combining standardized clinical examination, serum biomarkers, imaging and classically electrophysiological examinations, (among them auditive evoked potentials or AEP) but none has a sufficient sensitivity/specificity. In a preliminary study, the investigators developed an algorithm from the signal collected with AEP, and generated a probability map to visually classify the participants after the algorithm processing. Participants could be classified either with a good neurological prognosis or with bad neurological prognosis or death.

The investigators hypothesize that the "PRECOM" tool, applied blindly to a large prospective multicenter cohort of patients admitted to intensive care for coma in the aftermath of CA will predict neurological prognosis at 3 months with high sensitivity and specificity.

DETAILED DESCRIPTION:
Evaluating the prognosis of comatose participants after cardiac arrest (CA) in the intensive care unit remains challenging. It requires a multimodal approach combining standardized clinical examination, serum biomarkers, imaging and classically electrophysiological examinations: 1 / the electroencephalogram, bad prognosis assessed when the electroencephalogram (EEG) is discontinuous, areactive, monotone,…), 2 / somesthetic evoked potentials, the absence of the N20 cortical wave has a specificity of poor prognosis of 68-100% and 3 / auditory evoked potentials (AEP), the presence of mismatchnegativity (MMN) would be of good prognosis with a specificity up to 90% but rarely performed in current practice. Routinely, these examinations are sometimes difficult to interpret in sedated participants, in an intensive care unit environment that generates numerous artefacts. Above all, all these techniques require the presence of a neurophysiology unit, with few experts available.

In a preliminary study, in collaboration with the applied mathematics laboratory of the ENS (Ecole Normale Supérieure), an algorithm was developed from the signal extracted from AEP. A probability map was generated with a software allowing to visually classify the participants after processing signal by the algorithm in a cluster of points with a high specificity into "good neurological prognosis" and "bad neurological prognosis". Neither artifacts or sedation prevented data analysis.

The investigators hypothesize that the "PRECOM" tool, applied blindly to a large prospective multicenter cohort of participants admitted to intensive care for coma in the aftermath of a caridiac arrest will predict the neurological prognosis of participants with high sensitivity and specificity. This tool, carried out during the first week of the coma, will be compared to a standardized procedure used routinely by the participating resuscitators.

ELIGIBILITY:
Inclusion Criteria:

* Age above18 years old
* Patient affiliated to a French Heath Care Insurance
* Admitted in the intensive care unit (ICU) for coma post extra- or intra-hospital cardiac arrest (CA) with shockable or non-shockable rhythm
* Persistent coma on day 3 after post CA, defined by the inability to respond to a verbal command in an appropriate manner (motor Glasgow components ≤ 3) and at the time of neurophysiological recordings (D3-D7 ± week -end).

Exclusion Criteria:

* Decision to limit resuscitation therapies taken by the resuscitation team
* Inability to perform the auditory evoked potentials (AEP) (deafness, skin lesion or any condition preventing to record AEP).
* Opposition by the trusted person or by the patient once he/she wakes up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to intensive care following a cardica arrest.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-05-29 (Estimated)

PRIMARY OUTCOMES:
Awakening within 3 months | within 3 months ± 2 weeks after inclusion
  Awakening is defined as normal motor activity in response to the 3 instructions for the motor component M of the FOUR score (show your thumb, make the V for victory and show your fist; M = 4). This criterion will be collected by the doctor in charge of the patient at the time of the assessment and will be dated.

SECONDARY OUTCOMES:
CPC score within 3 months | 3 months ± 2 weeks after inclusion
  CPC (Cerebral Performance Category) score is performed wether patient is still hospitalized or returned home. It is performed by phone call if patient returned home.
  Range of values rates neurological status after cardiac arrest on a scale of 1 to 5 (1 for good cerebral performance up to 5 for brain death).
mRS score within 3 months | 3 months ± 2 weeks after inclusion
  mRS (Modified Rankin Scale) scores is performed wether patient is still hospitalized or returned home. It is performed by phone call if patient returned home.
  mRS (modified Rankin Scale) scale measures degree of disability/dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Score can be between 0 (no symptoms at all) and 5 (major disability : bedridden, incontinent and requiring constant nursing care and attention).
FOUR score within 3 months | 3 months ± 2 weeks after inclusion
  FOUR (Full Outline of UnResponsiveness) score is performed only if patient is still hospitalized (being awake or not).
  FOUR score is a grading scale for assessing the level of consciousness performed on patients with severe neurologic impairment..It addresses four domains of neurological functioning: Eye response; Motor response ; Brainstem score and Respiratory score.
  Score is ranging from 0 to 16 where the lower the score, the greater the coma gravity.
GOSE score within 3 months | 3 months ± 2 weeks after inclusion
  GOSE (Extended Glasgow Outcome Scale) score is performed wether patient is still hospitalized or returned home.
  GOSE score classifies global outcomes in traumatic brain injury survivors. It rates patient status into one of eight categories ranging from 8 (Upper good recovery) to 1 (Dead).
CPC score within 6 months | 6 months ± 2 weeks after inclusion
  CPC (Cerebral Performance Category) score is performed wether patient is still hospitalized or returned home. It is performed by phone call if patient returned home.
  Range of values rates neurological status after cardiac arrest on a scale of 1 to 5 (1 for good cerebral performance up to 5 for brain death).
mRS score within 6 months | within 6 months ± 2 weeks after inclusion
  mRS (Modified Rankin Scale) scores is performed wether patient is still hospitalized or returned home. It is performed by phone call if patient returned home.
  mRS (modified Rankin Scale) scale measures degree of disability/dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Score can be between 0 (no symptoms at all) and 5 (major disability : bedridden, incontinent and requiring constant nursing care and attention).
GOSE score within 6 months | within 6 months ± 2 weeks after inclusion
  GOSE (Extended Glasgow Outcome Scale) score is performed wether patient is still hospitalized or returned home.
  GOSE score classifies global outcomes in traumatic brain injury survivors. It rates patient status into one of eight categories ranging from 8 (Upper good recovery) to 1 (Dead).
Awakening within 6 months ± 2 weeks | within 6 months ± 2 weeks after inclusion
  Awakening is defined as normal motor activity in response to the 3 instructions for the motor component M of the FOUR score (show your thumb, make the V for victory and show your fist; M = 4). This criterion will be collected by the doctor in charge of the patient at the time of the assessment and will be dated. The measurement takes place only if patient is still hospitalized.
CRS-R score within 6 months | within 6 months ± 2 weeks after inclusion
  CRS-R (Coma Recovery Scale - Revised) is a standardized neurobehavioral assessment measure designed for use in patients with disorders of consciousness. The scale is intented to be used to establish diagnosis, monitor behavioral recovery and predict outcome. It is performed only if patient is still hospitalized.
  The total score ranges between 0 (worst) and 23 (best).
PRECOM tool - first week of coma | Inclusion visit (3 to 7 days after cardiac arrest +/- 2 days if week-end)
  Comparison of the ability of the PRECOM tool using clinical and electrophysiological data at inclusion (the first week of coma), to classify patients with good prognosis, poor prognosis and indeterminate prognosis with respect to this same categorization using the usual evaluation criteria performed routinely by participating resuscitations (clinical examination and EEG for all and evoked potentials in addition for some).
PRECOM tool - second week of coma | One week visit (one week after inclusion visit +/- 2 days)
  Comparison of the ability of the PRECOM tool using clinical and electrophysiological data the second week of coma, to classify patients with good prognosis, poor prognosis and indeterminate prognosis with respect to this same categorization using the usual evaluation criteria performed routinely by participating resuscitations (clinical examination and EEG for all and evoked potentials in addition for some).
PRECOM tool - first and second week of coma | Inclusion and one week visits
  Comparison of the ability of the PRECOM tool using combinaison of clinical and electrophysiological data collected both at inclusion and one week later (the first two weeks of coma), to classify patients with good prognosis, poor prognosis and indeterminate prognosis with respect to this same categorization using the usual evaluation criteria performed routinely by participating resuscitations (clinical examination and EEG for all and evoked potentials in addition for some).
Awakening - second week of coma | One week visit (one week after inclusion visit +/- 2 days)
  Awakening is defined as normal motor activity in response to the 3 instructions for the motor component M of the FOUR score (show your thumb, make the V for victory and show your fist; M = 4). This criterion will be collected by the doctor in charge of the patient at the time of the assessment and will be dated.
NSE blood marker | 3 days post cardiac arrest
  Comparison of the ability to predict awakening with the PRECOM tool using the NSE blood marker (neuron- spécific enolase) collected 3 days after cardiac arrest between the patients awakened from the coma and those who are not.
Glial blood markor | Inclusion visit (3 to 7 days after cardiac arrest +/- 2 days if week-end)
  Comparison of the ability to predict awakening with the PRECOM tool using the Glial Fibrillary Acidic Protein (GFAP) collected at the inclusion visit between the patients awakened from the coma and those who are not.
Neuronal blood markor | Inclusion visit (3 to 7 days after cardiac arrest +/- 2 days if week-end)
  Comparison of the ability to predict awakening with the PRECOM tool using the Neurofilament blood marker collected at the inclusion visit between the patients awakened from the coma and those who are not.
Inflammatory blood markor | Inclusion visit (3 to 7 days after cardiac arrest +/- 2 days if week-end)
  Comparison of the ability to predict awakening with the PRECOM tool using the inflammatory blood markers : Kynurenine and Tryptophan; collected at the inclusion visit between the patients awakened from the coma and those who are not.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie KUBIS, Md,PhD, Study Director — APHP Lariboisière Hospital, Clinical Physiology Department
Locations (7):
- France (7):
  - APHP Avicenne Hospital - Réanimation médico-chirurgicale, Bobigny
  - APHP Lariboisière Hospital, Clinical Physiology Department, Paris
  - APHP Laribosière Hospital - Service de Réanimation Médical et Toxicologique, Paris
  - APHP Cochin Hospital - médecine intensive-réanimation, Paris
  - APHP HEGP hospital - Réanimation médicale, Paris
  - APHP Bichat Hospital -Médecine intensive - réanimation infectieuse, Paris
  - Delafontaine Hospital - médecine intensive-réanimation, Saint-Denis

IPD SHARING:
Plan to Share IPD: No